CLINICAL TRIAL: NCT00005535
Title: Gene Mapping for Quantitative Traits
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5068; R01HL055976 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2002-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To conduct gene mapping studies for quantitative traits.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The study built upon existing sib-pair methods for multipoint mapping of Quantitative Trait Loci (QTL)s. It greatly expanded upon the statistical methodology to identify and localize QTLs for complex traits by merging sib-pair methods with a powerful twin design which used phenotypic data on monozygotic (identical) and dizygotic (fraternal) twins to resolve phenotypic variability into genetic and non-genetic components, and partition human quantitative genetic variation into effects due to loci on specific chromosomal regions. This quantitative methodology was applied to risk factors for cardiovascular disease -- one of the most pressing health problems in Western society. Population-based samples of Dutch, Swedish, and Australian twins had been identified in previous studies, phenotypic measures on lipids, lipoproteins, and other important cardiovascular risk factors had been obtained, and blood had been banked in a valuable resource which was available for use in this study. In 500 DZ twin pairs, a series of 175 highly polymorphic microsatellite markers were detected using an automated process for detecting fluorescent signals. These data were analyzed using the new statistical methods both to confirm the effects of a series of candidate loci and to test for the effects of previously unknown QTLs.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-09; Study Completion 2000-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Vogler — Penn State University

REFERENCES:
- [Background] Nelson TL, Vogler GP, Pedersen NL, Miles TP. Genetic and environmental influences on waist-to-hip ratio and waist circumference in an older Swedish twin population. Int J Obes Relat Metab Disord. 1999 May;23(5):449-55. doi: 10.1038/sj.ijo.0800840. PMID 10375046
- [Background] Vogler GP, Tang W, Nelson TL, Hofer SM, Grant JD, Tarantino LM, Fernandez JR. A multivariate model for the analysis of sibship covariance structure using marker information and multiple quantitative traits. Genet Epidemiol. 1997;14(6):921-6. doi: 10.1002/(SICI)1098-2272(1997)14:63.0.CO;2-N. PMID 9433601
- [Background] McClearn GE, Vogler GP. Genetics and behavioral medicine: the error of the error term. Behav Med. 1997 Winter;22(4):150-1. doi: 10.1080/08964289.1997.10543547. No abstract available. PMID 9138622
- [Background] Vogler GP, McClearn GE, Snieder H, Boomsma DI, Palmer R, de Knijff P, Slagboom PE. Genetics and behavioral medicine: risk factors for cardiovascular disease. Behav Med. 1997 Winter;22(4):141-9. doi: 10.1080/08964289.1997.10543546. PMID 9138621
- [Background] Beekman M, Lakenberg N, Cherny SS, de Knijff P, Kluft CC, van Ommen GJ, Vogler GP, Frants RR, Boomsma DI, Slagboom PE. A powerful and rapid approach to human genome scanning using small quantities of genomic DNA. Genet Res. 2001 Apr;77(2):129-34. doi: 10.1017/s001667230100492x. PMID 11355568
- [Background] Beekman M, Heijmans BT, Martin NG, Pedersen NL, Whitfield JB, DeFaire U, van Baal GC, Snieder H, Vogler GP, Slagboom PE, Boomsma DI. Heritabilities of apolipoprotein and lipid levels in three countries. Twin Res. 2002 Apr;5(2):87-97. doi: 10.1375/1369052022956. PMID 11931686